CLINICAL TRIAL: NCT03703297
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multi-center, International Study of Durvalumab or Durvalumab and Tremelimumab as Consolidation Treatment for Patients With Limited Stage Small Cell Lung Cancer Who Have Not Progressed Following Concurrent Chemoradiation Therapy (ADRIATIC)
Brief Title: Study of Durvalumab + Tremelimumab, Durvalumab, and Placebo in Limited Stage Small-Cell Lung Cancer in Patients Who Have Not Progressed Following Concurrent Chemoradiation Therapy
Acronym: ADRIATIC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D933QC00001; 2018-000867-10 (EudraCT Number)
Record Dates: First submitted 2018-09-19; First posted 2018-10-11 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; SCLC; LS-SCLC; Limited Stage; Carcinoma; Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma; Lung Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Durvalumab + Placebo (Experimental): Durvalumab monotherapy: Durvalumab (1500 mg intravenous [IV]) q4w in combination with placebo saline solution (IV) q4w for up to 4 doses/cycles each, followed by durvalumab 1500 mg q4w. The first durvalumab monotherapy 1500 mg dose q4w will be 4 weeks after the final dose of durvalumab in combination with placebo saline solution.
  Interventions: Drug: Durvalumab; Other: Placebo
- Durvalumab + Tremelimumab (Experimental): Durvalumab in combination with tremelimumab: Durvalumab (1500 mg IV) q4w in combination with tremelimumab (75 mg IV) q4w for up to 4 doses/cycles each, followed by durvalumab 1500 mg q4w. The first durvalumab monotherapy 1500 mg dose q4w will be 4 weeks after the final dose of durvalumab in combination with tremelimumab.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Placebo + Placebo (Placebo Comparator): Placebo: Placebo saline solution (IV) q4w in combination with a second placebo saline solution (IV) q4w for up to 4 doses/cycles each, followed by a single placebo saline solution q4w. The first placebo saline solution monotherapy dose q4w will be 4 weeks after the final dose of the 2 placebo saline solutions in combination.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous infusion)
  Other Names: MEDI4736
  Arms: Durvalumab + Placebo; Durvalumab + Tremelimumab
Drug: Tremelimumab — Tremelimumab IV (intravenous infusion)
  Arms: Durvalumab + Tremelimumab
Other: Placebo — Placebo IV (intravenous infusion)
  Arms: Durvalumab + Placebo; Placebo + Placebo

SUMMARY:
This is a Phase III, Randomized, Double-blind, Placebo-controlled, Multi-center, International Study of Durvalumab or Durvalumab and Tremelimumab as Consolidation Treatment for Patients with LS-SCLC Who Have Not Progressed Following Concurrent Chemoradiation Therapy

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically documented limited-stage small cell lung cancer (stage I-III).
2. Received 4 cycles of chemotherapy concurrent with radiotherapy, which must be completed within 1 to 42 days prior to randomization and the first dose of IP. Chemotherapy must contain platinum and IV etoposide. Radiotherapy must be either total 60-66 Gy over 6 weeks for the standard QD regimen or total 45 Gy over 3 weeks for hyperfractionated BD schedules.
3. PCI may be delivered at the discretion of investigator and local standard of care, and must be conducted after the end of cCRT and completed between 1 to 42 days to first dose of IP.

4 .Have not progressed following definitive concurrent chemoradiation 5 .Life expectancy ≥ 12 weeks at Day 1. 6. ECOG 0 or 1 at enrolment.

Exclusion criteria:

1. Extensive-stage SCLC
2. Active or prior documented autoimmune or inflammatory disorders
3. Uncontrolled intercurrent illness, including but not limited to interstitial lung disease.
4. Active infection including tuberculosis, HIV, hepatitis B and C
5. Patients who received sequential chemotherapy and radiotherapy (no overlap of RT with chemotherapy)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2026-10-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Haiyi Jiang, M.D., Study Director — AstraZeneca
Locations (159):
- United States (33):
  - Research Site, Tucson, Arizona
  - Research Site, Santa Rosa, California
  - Research Site, New Haven, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Orange City, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Hines, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Summit, New Jersey
  - Research Site, New Hyde Park, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Kennewick, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Huntington, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (5):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Rosario
- Belgium (5):
  - Research Site, Aalst
  - Research Site, Anderlecht
  - Research Site, Brussels
  - Research Site, Hasselt
  - Research Site, Roeselare
- Canada (8):
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, CA
  - Research Site, Winnipeg, Manitoba
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (15):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- Czechia (4):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
- Germany (11):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Heidelberg
  - Research Site, Mainz
  - Research Site, Münster
  - Research Site, Oldenburg
  - Research Site, Regensburg
  - Research Site, Stuttgart
  - Research Site, Würzburg
- India (2):
  - Research Site, Bengaluru
  - Research Site, Gūrgaon
- Italy (7):
  - Research Site, Brescia
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Terni
- Japan (16):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Iwakuni-shi
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Tokushima
  - Research Site, Ube-shi
- Netherlands (5):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Harderwijk
  - Research Site, Hengelo
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (7):
  - Research Site, Kazan'
  - Research Site, Kirov
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Ufa
  - Research Site, Volgograd
- South Korea (8):
  - Research Site, Changwon-si
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Jinju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (8):
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
  - Research Site, Yunlin
- Turkey (Türkiye) (8):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Konya
  - Research Site, Samsun
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Truro
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Zenke Y, Shiraishi Y, Goto Y, Azuma K, Okishio K, Ogino H, Horio Y, Oizumi S, Hayama M, Nii M, Harada M, Mann H, Olivo YS, Jiang H, Senan S. Durvalumab Post Concurrent Chemoradiotherapy in Japanese Patients With Limited-Stage Small-Cell Lung Cancer in the Phase 3 ADRIATIC Trial. Cancer Sci. 2025 Nov;116(11):3171-3184. doi: 10.1111/cas.70188. Epub 2025 Sep 21. PMID 40976711
- [Derived] Cheng Y, Spigel DR, Cho BC, Laktionov KK, Fang J, Chen Y, Zenke Y, Lee KH, Wang Q, Navarro A, Bernabe R, Buchmeier EL, Chang JW, Shiraishi Y, Sezgin Goksu S, Badzio A, Shi A, Daniel DB, Hoa NTT, Zemanova M, Mann H, Gowda H, Jiang H, Senan S; ADRIATIC Investigators. Durvalumab after Chemoradiotherapy in Limited-Stage Small-Cell Lung Cancer. N Engl J Med. 2024 Oct 10;391(14):1313-1327. doi: 10.1056/NEJMoa2404873. Epub 2024 Sep 13. PMID 39268857
- [Derived] Senan S, Okamoto I, Lee GW, Chen Y, Niho S, Mak G, Yao W, Shire N, Jiang H, Cho BC. Design and Rationale for a Phase III, Randomized, Placebo-controlled Trial of Durvalumab With or Without Tremelimumab After Concurrent Chemoradiotherapy for Patients With Limited-stage Small-cell Lung Cancer: The ADRIATIC Study. Clin Lung Cancer. 2020 Mar;21(2):e84-e88. doi: 10.1016/j.cllc.2019.12.006. Epub 2019 Dec 28. PMID 31948903
- See also: d933qc00001-csp-v5_for redaction_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933QC00001&attachmentIdentifier=3f92618b-645a-46cb-b59f-0d74a735a2ce&fileName=d933qc00001-csp-v5_for_redaction_Redacted.pdf&versionIdentifier=
- See also: d933qc00001-csp-v1-addendum-eu_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933QC00001&attachmentIdentifier=3f226cd4-d1d6-4641-8c9e-6f5ad1dc54c5&fileName=d933qc00001-csp-v1-addendum-eu_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933QC00001&attachmentIdentifier=95aa7044-7fca-47aa-933d-fa972ad5963b&fileName=d933qc00001-sap-ed-5_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933QC00001&attachmentIdentifier=72ddfb20-d1e8-46e1-b0fc-4ac97e3b7149&fileName=d933qc00001-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, double-blind, placebo-controlled trial studied participants with limited stage small-cell lung cancer who had not progressed after concurrent chemoradiation therapy at 164 sites in 19 countries. Interim results are based on data cut-off (DCO) date of 15 January 2024. 730 participants were randomized; the first 600 in a 1:1:1 ratio to durvalumab monotherapy (D), durvalumab plus tremelimumab combination therapy (D+T) or placebo (P), the remaining in a 1:1 ratio to D or P.
Pre-assignment Details: Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded independent data monitoring committee [IDMC]), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis.
Groups:
- Durvalumab: Participants received durvalumab monotherapy (1500 milligram [mg] for participants >30 kilogram [kg] in weight and a weight-based dosing equivalent to 20 mg/kg for participants <=30 kg in weight) via intravenous (IV) infusion once every 4 weeks (q4w), until clinical/Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)-defined radiological progression, intolerable toxicity, or for a maximum of 24 months, whichever occurred first.
- Durvalumab Plus Tremelimumab: Participants received durvalumab in combination with tremelimumab (1500 mg durvalumab in combination with 75 mg tremelimumab for participants >30 kg in weight and a weight-based dosing equivalent to 20 mg/kg durvalumab in combination with 1 mg/kg tremelimumab for participants <=30 kg in weight) via IV infusion once q4w, until clinical/RECIST 1.1-defined radiological progression, intolerable toxicity, or for a maximum of 24 months, whichever occurred first.
- Placebo: Participants received matching placebo via IV infusion once q4w for 4 doses/cycles each, until clinical/RECIST 1.1-defined radiological progression, intolerable toxicity, or for a maximum of 24 months, whichever occurred first.
Period: Overall Study
Arm/Group | Durvalumab | Durvalumab Plus Tremelimumab | Placebo
Started | 264 | 200 | 266
Safety Population | 262 | 0 | 265
Completed | 0 | 0 | 0
Not Completed | 264 | 200 | 266
Not completed — Death | 115 | 0 | 144
Not completed — Withdrawal by Subject | 9 | 0 | 11
Not completed — Ongoing at the time of DCO | 140 | 200 | 111

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants.
Groups:
- Durvalumab: Participants received durvalumab monotherapy (1500 mg for participants >30 kg in weight and a weight-based dosing equivalent to 20 mg/kg for participants <=30 kg in weight) via IV infusion once q4w, until clinical/RECIST 1.1-defined radiological progression, intolerable toxicity, or for a maximum of 24 months, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Durvalumab | Durvalumab Plus Tremelimumab | Placebo | Total
Number analyzed (Participants) | 264 | 200 | 266 | 730
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 160 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 162 | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | 104 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 104 | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 78 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 178 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 188 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 130 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 137 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | 1 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | 131 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 121 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Other | 2 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 5 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 14 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | 255 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 249 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Missing | 1 | NA — Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis. | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Durvalumab Versus Placebo: Progression-Free Survival (PFS) Assessed by Blinded Independent Central Review (BICR) Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: PFS per RECIST 1.1 assessed by BICR was defined as the time from the date of randomization until the date of objective disease progression (PD) or death (by any cause in the absence of progression) regardless of whether the participant withdrew from therapy or received another anticancer therapy prior to progression. PD was defined as at least a 20% increase in the sum of diameters of target lesions (TLs), taking as reference the smallest previous sum of diameters (nadir) - this included the baseline sum if that was the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm) from nadir. Median PFS was calculated using Kaplan-Meier method and its confidence interval (CI) using Brookmeyer-Crowley method.
Time Frame: Response evaluations performed every 8 weeks (q8w) ± 1 week up to 72 weeks, then every 12 weeks (q12w) ± 1 week up to 96 weeks, and then every 24 weeks (q24w) thereafter until PD, up to DCO date 15 January 2024 (a maximum of approximately 1936 days)
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 264 | 266
months | 16.6 [10.2 to 28.2] | 9.2 [7.4 to 12.9]
Statistical Analysis 1: Comparison: Durvalumab vs Placebo; Test type: Superiority; p = 0.01608, Log Rank; The analysis was performed using the stratified log-rank test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.606 to 0.950] — Hazard ratio and CI calculated using stratified Cox proportional hazards model,adjusting for tumor,node and metastasis(TNM) stage, receipt of prophylactic cranial irradiation(PCI),with treatment as only covariate and ties handled by Efron approach

2. Primary Outcome: Durvalumab Versus Placebo: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until death due to any cause. Median OS was calculated using Kaplan-Meier method and its CI using Brookmeyer-Crowley method.
Time Frame: From date of randomization until death due to any cause, up to DCO date 15 January 2024 (a maximum of approximately 1936 days)
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 264 | 266
months | 55.9 [37.3 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at the DCO. | 33.4 [25.5 to 39.9]
Statistical Analysis 1: Comparison: Durvalumab vs Placebo; Test type: Superiority; p = 0.01042, Log Rank; The analysis was performed using the stratified log-rank test; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.569 to 0.928] — Hazard ratio and CI were calculated using stratified Cox proportional hazards model, adjusting for receipt of PCI, with treatment as only covariate and ties handled by Efron approach

3. Secondary Outcome: Durvalumab Plus Tremelimumab Combination Versus Placebo: Progression-Free Survival Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: PFS per RECIST 1.1 assessed by BICR is defined as the time from the date of randomization until the date of objective PD or death (by any cause in the absence of progression) regardless of whether the participant withdraws from therapy or receives another anticancer therapy prior to progression. PD is defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir) - this includes the baseline sum if that is the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm from nadir.
Time Frame: Response evaluations performed q8w ± 1 week up to 72 weeks, then q12w ± 1 week up to 96 weeks, and then q24w thereafter until PD, up to approximately 89 months
Reporting Status: Not Posted, anticipated posting 2027-03

4. Secondary Outcome: Durvalumab Plus Tremelimumab Combination Versus Placebo: Overall Survival
Description: OS is defined as the time from the date of randomization until death due to any cause.
Time Frame: From date of randomization until death due to any cause, up to approximately 89 months
Reporting Status: Not Posted, anticipated posting 2027-03

5. Secondary Outcome: Durvalumab Versus Placebo: Objective Response Rate (ORR) Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: ORR per RECIST 1.1 assessed by BICR was defined as the percentage of participants with at least 1 visit response of complete response (CR) or partial response (PR) (i.e., unconfirmed response). CR was defined as disappearance of all TLs since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to <10 mm. PR was defined as at least a 30% decrease in the sum of the diameters of TL, taking as reference the baseline sum of diameters.
Time Frame: Response evaluations performed q8w ± 1 week up to 72 weeks, then q12w ± 1 week up to 96 weeks, and then q24w thereafter until PD, up to DCO date 15 January 2024 (a maximum of approximately 1936 days)
Population: The FAS included all randomized participants. Only participants with measurable disease at baseline per BICR are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 175 | 169
percentage of participants | 30.3 | 32.0

6. Secondary Outcome: Durvalumab Plus Tremelimumab Combination Versus Placebo: Objective Response Rate Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: ORR per RECIST 1.1 assessed by BICR is defined as the percentage of participants with at least 1 visit response of CR or PR (i.e., unconfirmed response). CR is defined as disappearance of all TLs since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to <10 mm. PR is defined as at least a 30% decrease in the sum of the diameters of TL, taking as reference the baseline sum of diameters.
Time Frame: From date of randomization until death due to any cause, up to approximately 89 months
Reporting Status: Not Posted, anticipated posting 2027-03

7. Secondary Outcome: Durvalumab Versus Placebo: Percentage of Participants Progression-Free at 18 Months Following Randomization (PFS18) Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: PFS per RECIST 1.1 assessed by BICR was defined as the time from the date of randomization until the date of objective PD or death (by any cause in the absence of progression) regardless of whether the participant withdrew from therapy or received another anticancer therapy prior to progression. PD was defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir) - this included the baseline sum if that was the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm from nadir. The PFS18 was defined as the Kaplan-Meier estimate of PFS per RECIST 1.1 as assessed by BICR at 18 months following randomization.
Time Frame: Month 18
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 264 | 266
percentage of participants | 48.8 [42.2 to 55.0] | 36.1 [29.9 to 42.2]

8. Secondary Outcome: Durvalumab Plus Tremelimumab Combination Versus Placebo: Percentage of Participants Progression-Free at 18 Months Following Randomization Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: PFS per RECIST 1.1 assessed by BICR is defined as the time from the date of randomization until the date of objective PD or death (by any cause in the absence of progression) regardless of whether the participant withdraws from therapy or receives another anticancer therapy prior to progression. PD is defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir) - this includes the baseline sum if that is the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm from nadir. The PFS18 is defined as the Kaplan-Meier estimate of PFS per RECIST 1.1 as assessed by BICR at 18 months following randomization.
Time Frame: Month 18
Reporting Status: Not Posted, anticipated posting 2027-03

9. Secondary Outcome: Durvalumab Versus Placebo: Percentage of Participants Progression-Free at 24 Months Following Randomization (PFS24) Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: PFS per RECIST 1.1 assessed by BICR was defined as the time from the date of randomization until the date of objective PD or death (by any cause in the absence of progression) regardless of whether the participant withdrew from therapy or received another anticancer therapy prior to progression. PD was defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir) - this included the baseline sum if that was the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm from nadir. The PFS24 was defined as the Kaplan-Meier estimate of PFS per RECIST 1.1 as assessed by BICR at 24 months following randomization.
Time Frame: Month 24
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 264 | 266
percentage of participants | 46.2 [39.6 to 52.5] | 34.2 [28.2 to 40.3]

10. Secondary Outcome: Durvalumab Plus Tremelimumab Combination Versus Placebo: Percentage of Participants Progression-Free at 24 Months Following Randomization Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: PFS per RECIST 1.1 assessed by BICR is defined as the time from the date of randomization until the date of objective PD or death (by any cause in the absence of progression) regardless of whether the participant withdraws from therapy or receives another anticancer therapy prior to progression. PD is defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir) - this included the baseline sum if that is the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm from nadir. The PFS24 is defined as the Kaplan-Meier estimate of PFS per RECIST 1.1 as assessed by BICR at 24 months following randomization.
Time Frame: Month 24
Reporting Status: Not Posted, anticipated posting 2027-03

11. Secondary Outcome: Durvalumab Plus Tremelimumab Combination Versus Placebo: Time to Death or Distant Metastasis (TTDM) Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: TTDM per RECIST 1.1 is defined as the time from the date of randomization until the first date of distant metastasis or death in the absence of distant metastasis. Distant metastasis is defined as any new lesion that is outside of the radiation field according to RECIST 1.1 or proven by biopsy.
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2027-03

12. Secondary Outcome: Durvalumab Versus Placebo: Percentage of Participants Alive at 24 Months From Randomization (OS24)
Description: OS was defined as the time from the date of randomization until death due to any cause. The OS24 was defined as the Kaplan-Meier estimate of OS at 24 months after randomization.
Time Frame: Month 24
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 264 | 266
percentage of participants | 68.0 [61.9 to 73.3] | 58.5 [52.3 to 64.3]

13. Secondary Outcome: Durvalumab Plus Tremelimumab Combination Versus Placebo: Percentage of Participants Alive at 24 Months From Randomization
Description: OS is defined as the time from the date of randomization until death due to any cause. The OS24 is defined as the Kaplan-Meier estimate of OS at 24 months after randomization.
Time Frame: Month 24
Reporting Status: Not Posted, anticipated posting 2027-03

14. Secondary Outcome: Durvalumab Versus Placebo: Percentage of Participants Alive at 36 Months From Randomization (OS36)
Description: OS was defined as the time from the date of randomization until death due to any cause. The OS36 was defined as the Kaplan-Meier estimate of OS at 36 months after randomization.
Time Frame: Month 36
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Placebo
Number analyzed (Participants) | 264 | 266
percentage of participants | 56.5 [50.0 to 62.5] | 47.6 [41.3 to 53.7]

15. Secondary Outcome: Durvalumab Plus Tremelimumab Combination Versus Placebo: Percentage of Participants Alive at 36 Months From Randomization
Description: OS is defined as the time from the date of randomization until death due to any cause. The OS36 is defined as the Kaplan-Meier estimate of OS at 36 months after randomization.
Time Frame: Month 36
Reporting Status: Not Posted, anticipated posting 2027-03

16. Secondary Outcome: Durvalumab Plus Tremelimumab Combination Versus Placebo: Time From Randomization to Second Progression (PFS2)
Description: PFS2 is defined as the time from the date of randomization to the earliest of the progression event subsequent to the first subsequent anticancer therapy (excluding radiotherapy) or death. The date of second progression is recorded by the Investigator in the eCRF at each assessment and defined according to local standard clinical practice and might involve any of the following: objective radiological imaging, symptomatic progression, or death.
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2027-03

17. Secondary Outcome: Durvalumab Versus Durvalumab Plus Tremelimumab: Progression-Free Survival Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: as for outcome 3
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2027-03

18. Secondary Outcome: Durvalumab Versus Durvalumab Plus Tremelimumab: Objective Response Rate Assessed by Blinded Independent Central Review Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: as for outcome 6
Time Frame: From date of randomization until death due to any cause, up to approximately 89 months
Reporting Status: Not Posted, anticipated posting 2027-03

19. Secondary Outcome: Durvalumab Versus Durvalumab Plus Tremelimumab: Overall Survival
Description: OS is defined as the time from the date of randomization until death due to any cause.
Time Frame: From date of randomization until death due to any cause, up to approximately 89 months
Reporting Status: Not Posted, anticipated posting 2027-03

20. Secondary Outcome: Durvalumab Plus Tremelimumab Versus Placebo: Change From Baseline in Patient-Reported Symptoms as Assessed by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires (EORTC QLQ)
Description: Patient-reported outcomes for 5 disease related symptoms will be assessed using EORTC QLQ-Core 30 (C30) items questionnaire (fatigue, appetite loss) and EORTC QLQ-Lung Cancer module 13 (LC13) (dyspnea, cough and pain in chest). An outcome variable consisting of a score from 0 to 100 will be derived for each of the symptom scales/symptom items, functional scales, and global health status (GHS) scale with higher scores on GHS/QoL and functioning scales representing better health status/function, but higher scores on symptom scales/items representing greater symptom severity.
Time Frame: Baseline (Day 1) and up to approximately 89 months
Reporting Status: Not Posted, anticipated posting 2027-03

21. Secondary Outcome: Durvalumab: Serum Concentration of Durvalumab
Description: Blood samples were collected to determine the concentration of durvalumab.
Time Frame: End of infusion on Cycle 1 Day 1, pre-infusion on Cycle 2 (Week 4), Cycle 5 (Week 16) and Cycle 26 (Week 100) and Month 3 post last dose of study treatment (Week 119) (each treatment cycle is 28 days)
Population: The pharmacokinetic (PK) population included all participants who received at least 1 dose of study drug per the protocol for whom any post-dose data were available and who did not violate or deviate from the protocol in ways that would have significantly affected the PK analyses. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Durvalumab
Number analyzed (Participants) | 222
microgram per milliliter (mcg/mL)
  Cycle 1 Day 1: End of infusion | 431.00 (327.861)
  Cycle 2 (Week 4): Pre-infusion: number analyzed (Participants) | 215
  Cycle 2 (Week 4): Pre-infusion | 89.57 (107.228)
  Cycle 5 (Week 16): Pre-infusion: number analyzed (Participants) | 119
  Cycle 5 (Week 16): Pre-infusion | 159.63 (58.561)
  Cycle 26 (Week 100): Pre-infusion: number analyzed (Participants) | 46
  Cycle 26 (Week 100): Pre-infusion | 178.20 (65.422)
  Month 3 follow-up: number analyzed (Participants) | 118
  Month 3 follow-up | 44.97 (36.026)

22. Secondary Outcome: Durvalumab Plus Tremelimumab: Serum Concentration of Tremelimumab
Description: Blood samples will be collected to determine the concentration of tremelimumab.
Time Frame: Up to approximately 27 months
Reporting Status: Not Posted, anticipated posting 2027-03

23. Secondary Outcome: Durvalumab: Number of Participants With Anti-Drug Antibody (ADA) Response to Durvalumab
Description: Blood samples were collected to determine the presence of ADAs for durvalumab using validated assays. Treatment-emergent ADA-positive was defined as either treatment-induced (post-baseline ADA-positive only) or treatment-boosted ADA (baseline positive ADA titer that was boosted to ≥4 fold during the study period). Treatment-induced ADA was defined as ADA positive post-baseline and not detected at baseline. Treatment-boosted ADA was defined as a baseline positive ADA titer that was boosted to a 4-fold or higher level (greater than the analytical variance of the assay) following drug administration. Number of participants with treatment-emergent ADA (ADA incidence) are presented.
Time Frame: From first dose of study drug (Day 1) up to DCO date 15 January 2024 (a maximum of approximately 1936 days)
Population: The ADA population included all participants in the safety analysis set who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 206
Participants | 7

24. Secondary Outcome: Durvalumab Plus Tremelimumab: Number of Participants With Anti-Drug Antibody (ADA) Response to Tremelimumab
Description: Blood samples will be collected to determine the presence of ADAs for tremelimumab using validated assays. Treatment-emergent ADA-positive is defined as either treatment-induced (post-baseline ADA-positive only) or treatment-boosted ADA (baseline positive ADA titer that was boosted to ≥4 fold during the study period). Treatment-boosted ADA is defined as a baseline positive ADA titer that was boosted to a 4-fold or higher level (greater than the analytical variance of the assay) following drug administration. Treatment-induced ADA is defined as ADA positive post-baseline and not detected at baseline.
Time Frame: Up to approximately 30 months
Reporting Status: Not Posted, anticipated posting 2027-03

25. Secondary Outcome: Durvalumab Versus Durvalumab Plus Tremelimumab: Number of Participants With Positive Programmed Death Ligand 1 (PD-L1) Status Based on Progression-Free Survival, Overall Survival, and Objective Response Rate
Description: Blood samples will be collected for clinical biomarker testing and a tumor specimen will be collected as per tumor specimen collection requirements. The specimen will be evaluated by immunohistochemistry to determine the expression of tumor specific antigens and immune markers. The PD-L1 is a biomarker and will be assessed using the VENTANA PD-L1 (SP263) assay.
Time Frame: Up to approximately 89 months
Reporting Status: Not Posted, anticipated posting 2027-03

ADVERSE EVENTS:
Time Frame: From first dose of study drug(Day 1)upto DCO date 15 January 2024(maximum of approximately 1936 days).Safety population:all participants who received at least 1 dose of study drug.Based on results of secondary objectives at interim analysis(reviewed by unblinded IDMC),data for D+T arm were to remain blinded to Sponsor as pre-specified in study's unblinding plan.Since D+T arm was blinded at time of posting results from this interim analysis,results for that arm will be posted at final analysis.
Description: All-cause mortality was assessed for FAS. 1 participant randomized to Durvalumab arm received 2 cycles of tremelimumab and in accordance with SAP was therefore not included in Durva or placebo safety population; will be included in D+T safety population when D+T arm is unblinded.
Arm/Group | Durvalumab | Durvalumab Plus Tremelimumab | Placebo
All-Cause Mortality (participants affected / at risk) | 115/264 | 0/0 | 146/266
Serious Adverse Events (participants affected / at risk) | 78/262 | 0/0 | 64/265
Other Adverse Events (participants affected / at risk) | 209/262 | 0/0 | 196/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=262) | Durvalumab Plus Tremelimumab (N=0) | Placebo (N=265)
Gastritis (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | NA | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | NA | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | NA | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | NA | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | NA | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | NA | 1 (1)
Asthenia (General disorders) | 0 (0) | NA | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | NA | 0 (0)
Device related thrombosis (General disorders) | 1 (1) | NA | 0 (0)
Fatigue (General disorders) | 1 (1) | NA | 1 (1)
Hernia (General disorders) | 1 (1) | NA | 0 (0)
Pyrexia (General disorders) | 0 (0) | NA | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | NA | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | NA | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | NA | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | NA | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | NA | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | NA | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | NA | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | NA | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | NA | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | NA | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | NA | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | NA | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | NA | 1 (1)
Empyema (Infections and infestations) | 0 (0) | NA | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | NA | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | NA | 1 (1)
Infection (Infections and infestations) | 0 (0) | NA | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | NA | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | NA | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | NA | 1 (1)
Pneumonia (Infections and infestations) | 12 (12) | NA | 10 (11)
Pneumonia bacterial (Infections and infestations) | 3 (3) | NA | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | NA | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | NA | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | NA | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | NA | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | NA | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | NA | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | NA | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | NA | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | NA | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | NA | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | NA | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | NA | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | NA | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | NA | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 13 (13) | NA | 7 (7)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | NA | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | NA | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | NA | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | NA | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | NA | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | NA | 0 (0)
Weight decreased (Investigations) | 1 (1) | NA | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | NA | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | NA | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | NA | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | NA | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | NA | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | NA | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | NA | 1 (1)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | NA | 1 (1)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | NA | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | NA | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | NA | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | NA | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | NA | 1 (1)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | NA | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | NA | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | NA | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | NA | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | NA | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | NA | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | NA | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | NA | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | NA | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | NA | 0 (0)
Device dislocation (Product Issues) | 0 (0) | NA | 1 (1)
Alcoholic psychosis (Psychiatric disorders) | 1 (1) | NA | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | NA | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | NA | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | NA | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | NA | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | NA | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | NA | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | NA | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | NA | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | NA | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | NA | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | NA | 1 (1)
Iliac artery stenosis (Vascular disorders) | 0 (0) | NA | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | NA | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | NA | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1) | NA | 0 (0)
Cataract (Eye disorders) | 1 (1) | NA | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | NA | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | NA | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | NA | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=262) | Durvalumab Plus Tremelimumab (N=0) | Placebo (N=265)
Nausea (Gastrointestinal disorders) | 33 (39) | NA | 29 (35)
Vomiting (Gastrointestinal disorders) | 12 (14) | NA | 17 (18)
Asthenia (General disorders) | 26 (32) | NA | 17 (18)
Fatigue (General disorders) | 31 (37) | NA | 33 (35)
COVID-19 (Infections and infestations) | 18 (18) | NA | 16 (16)
Anaemia (Blood and lymphatic system disorders) | 21 (28) | NA | 16 (19)
Pneumonia (Infections and infestations) | 19 (23) | NA | 11 (11)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 49 (51) | NA | 55 (57)
Alanine aminotransferase increased (Investigations) | 15 (22) | NA | 13 (19)
Weight decreased (Investigations) | 18 (20) | NA | 11 (17)
White blood cell count decreased (Investigations) | 18 (36) | NA | 11 (27)
Decreased appetite (Metabolism and nutrition disorders) | 44 (56) | NA | 34 (34)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (23) | NA | 29 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (16) | NA | 20 (23)
Dizziness (Nervous system disorders) | 32 (34) | NA | 20 (23)
Headache (Nervous system disorders) | 24 (26) | NA | 35 (38)
Insomnia (Psychiatric disorders) | 16 (16) | NA | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (44) | NA | 32 (38)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (27) | NA | 18 (22)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 20 (22) | NA | 10 (10)
Hyperthyroidism (Endocrine disorders) | 27 (29) | NA | 4 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 34 (39) | NA | 19 (19)
Rash (Skin and subcutaneous tissue disorders) | 28 (37) | NA | 16 (20)
Hypothyroidism (Endocrine disorders) | 42 (54) | NA | 10 (10)
Constipation (Gastrointestinal disorders) | 26 (30) | NA | 26 (28)
Diarrhoea (Gastrointestinal disorders) | 27 (28) | NA | 22 (32)

LIMITATIONS AND CAVEATS:
Based on the results of the secondary objectives at the interim analysis (reviewed by an unblinded IDMC), data for the D+T arm were to remain blinded to the Sponsor as pre-specified in the study's unblinding plan. Since the D+T arm was blinded at the time of posting the results from this interim analysis, results for that arm will be posted at the time of final analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03703297/Prot_003.pdf
  • Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT03703297/SAP_004.pdf